CLINICAL TRIAL: NCT04782635
Title: Effect of Artificial Intelligence on Nutritional Status of Children Post Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Shifa Trust Eye Hospital (Other)
Responsible Party: Principal Investigator, Maryam Zahid, Principal Investigator, Al-Shifa Trust Eye Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: AlShifaTrustEye
Record Dates: First submitted 2021-02-24; First posted 2021-03-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Post-cardiac Surgery

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI group (Experimental): * Care givers will be selected through permuted block.
  * They will be explained the procedure of intervention and written consent will be asked.
  * Mobile application will be installed in their mobile.
  * They will be explained the working of mobile application
  * Application will make a standard diet plan for the child according to the requirements of the child
  * Then the child will use the application for one month.
  * After one month patient will visit the doctor for routine checkup, during the visit patient will be asked for the usefulness of the application.
  * Nutritional status of the patient will be monitored including weight, height, clinical signs, dietary history and will be updated in application.
  * Then patient will follow the application for one month
  * After another one month patient will visit the doctor for routine checkup, during the visit patient will be asked for the usefulness of the application and nutritional status will be measured
  Interventions: Device: mobile based application
- usual care group (Other): * Caregivers (Mothers/fathers/guardians) will be selected through permuted block.
  * Patient weight, height, clinical signs will be noted.
  * Caregivers will be handed over pamphlet regarding dietary instructions on discharge.
  * After one month patient will visit the doctor for routine checkup, during the visit nutritional status of the patient will be checked and noted including weight, height, clinical signs and dietary history.
  * Patient will leave hospital with no added dietary instruction.
  * After one month patient will visit the doctor for routine checkup, during the visit nutritional status of the patient will be checked and noted weight, height, clinical sign, and dietary history.
  Interventions: Behavioral: Pamphlet

INTERVENTIONS:
Device: mobile based application — Application basic function would be support and improve nutrition status of children. Personalization of goals and challenges, daily intake of calories, carbohydrates, proteins, fats, minerals and vitamins will be tracked, food logging, food tracking, meal and supplement reminders, recipes, visual cues (remaining calories) will be notified, episodes of vomiting, meals missed, diarrhea, nausea will be recorded , meal planned according to the food preferences of child, food composition table, nutrition blogs and articles
  Arms: AI group
Behavioral: Pamphlet — A pamphlet which will be provide knowledge to the patients
  Arms: usual care group

SUMMARY:
The objective of the study will be to assess the effect of artificial intelligence on nutritional status of children post cardiac surgery in comparison to usual care group.To assess usefulness of diet related mobile application in comparison to usual care group.To identify diet related problems among children post cardiac surgery in both groups (usual care group and intervention group ).

DETAILED DESCRIPTION:
Research question Is there any impact of artificial intelligence on nutritional status of children post cardiac surgery?

Null hypothesis:

There is no impact of artificial intelligence on nutritional status of children post cardiac surgery

Operational definition:

1. Cardiac surgery There are large number of different surgical procedures (more than 150) in congenital heart disease, it became necessary the grouping into categories or relatively homogeneous strata, so that the comparisons between the outcomes were performed. The RACHS-1 method was developed by the Children's Hospital Boston team through a panel of 11 nationally representative members of pediatric cardiologists and cardiac surgeon. It allocated 207 surgical procedures in 6 different categories with similar risk for hospital mortality.
2. Artificial intelligence (AI) Artificial intelligence is a way to make machines think and behave intelligently. These machines are controlled by software inside them, so AI has a lot to do with intelligent software programs that can control these machines. It is a science that can help machines understand the world and accordingly react to situations in the same way the humans do.27
3. Nutritional status The state of a person's health in terms of the nutrients in his or her diet. Nutritional status assessment is the interpretation of anthropometric (using Length-for-age and Weight-for-age clinical growth charts and Z score), clinical (muscle dystrophy) and dietary data (food frequency table, usual dietary intake and mobile based application) to determine whether a person or groups of people are well nourished or malnourished.
4. Nutrition related mobile application Application basic function would be support and improve nutrition status of children. Personalization of goals and challenges, daily intake of calories, carbohydrates, proteins, fats, minerals and vitamins will be tracked, food logging, food tracking, meal and supplement reminders, recipes, visual cues (remaining calories) will be notified, episodes of vomiting, meals missed, diarrhea, nausea will be recorded , meal planned according to the food preferences of child, food composition table, nutrition blogs and articles

Material and Methods:

STUDY DESIGN:

Randomized controlled trial

SETTING:

Tertiary Care Cardiac hospital, Rawalpindi , Pakistan.

SAMPLING TECNIQUE:

Permuted block BLINDING Double blinded study

SAMPLE SIZE:

Sample size is estimated to be 96, 48 in each group i.e. intervention and control group

DATA ANALYSIS PROCEDURE All data will be analyzed using SPSS 23 Descriptive statistics

* Percentages and frequencies for all categorical variables
* Categorical Data will be presented in form of bar and chart
* Mean and standard deviation for continuous data. Inferential statistics
* For comparison of characteristics of patients between usual care group and intervention group:
* Independent t-test for continuous variables
* Chi square for categorical variables
* Pre-test and post-test difference in mean changes will be assessed by Split-plot ANOVA
* To compare outcomes between usual care group and intervention group Chi square group will be used

Ethical consideration The study will start after presenting research proposal and obtaining ethical approval from Ethical Review Committee of Pakistan Institute of Ophthalmology, Al-Shifa School of Public Health. A formal letter will be used that will include the information relevant to the study e.g., the purpose and duration of this study, the level of privacy and confidentiality of information with anonymity of the respondents. While conducting this study, informed consent from all participants will be taken verbally and in written form. Participation will be voluntary and individuals will be informed that they can withdraw at any time and that all data will be treated confidentially. Subjects will be assured of anonymity and confidentiality. Patients will be given a broad outline of the research, an indication of the type of information that is required, the reasons why the research is being carried out and how the information which they provided will be used.

Independent variable

1. Name
2. Gender
3. Age (months )
4. Ethnicity
5. Weight (lbs)
6. Height (cm)
7. Percentile (Weight for age )
8. Z score (weight for age )
9. Phone No:
10. Address
11. Education level of mother father
12. Smart phone knowledge (low/medium/high)
13. Monthly income
14. No of siblings
15. No. of family members
16. No of smart phones at home
17. Diagnosis
18. Primary surgery
19. RACH score (class 1/class 2)
20. CVA yes/no
21. Creatinine ________
22. Hb ________
23. Albumin level _______
24. Number of days in hospital
25. Number of days in ICU
26. Ventilator time
27. Reopened yes/ no
28. Food allergy Wheat ________ Milk __________ Nuts __________ Eggs___________ Other ___________
29. Anorexia yes/ no
30. Muscle dystrophy yes/ no
31. Calories required
32. Proteins required
33. Carbohydrates required
34. Fats required
35. All vitamins will be listed (required)
36. All minerals will be listed (required)

ELIGIBILITY:
Inclusion Criteria:

* Children of age 2-12 (early and middle childhood) years will be included in the study.
* Surgeries within first and second class of RACHS score are included in the study.
* Patients with smart phones and internet facilities are included in the study.
* Patients with caregivers who can read English are included in the study
* Patients discharged from the hospital will be selected

Exclusion Criteria:

* Patients with multiple congenital abnormalities and surgeries without an RACHS score are excluded.
* Patient who will be rehospitalized will be excluded from the research

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 61 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-03 (Actual)

PRIMARY OUTCOMES:
Weight changes | 2 months
  observe the Weight changes , weight for age , Z score weight for age in both groups
Caloric intake | 2 months
  Check the average calories intake consumed in both groups
Proteins intake | 2 months
  Check the average proteins consumed in both groups
Mobile application usage | 2 months
  Patients will be asked whether the language used in application on a likert scale ranging from very easy to very difficult , handling application will be ranging from very easy to very difficult, cost effectiveness will be ranging from yes to very costly, Visual cues in application will be ranged from useful to difficult to understand, Recipes in application will be ranged from being Useful to not useful, Meal reminders will be ranged from being useful to irritating
nutritional issues | 2 months
  Patient will be inquired regarding the episodes of vomiting, diarrhea, loss of appetite and other nutritional related problems

SECONDARY OUTCOMES:
carbohydrates intake | 2 months
  Measure average carbohydrates consumed in both groups (intervention and usual care group) in mg
fats intake | 2 months
  Measure average fats consumed in both groups (intervention and usual care group) in mg
Vitamins intake | 2 months
  Measure average vitamins consumed in both groups (intervention and usual care group) in mg and µg
Minerals intake | 2 months
  Measure average minerals consumed in both groups (intervention and usual care group) in mg and µg

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Armed Forces Institute of Cardiology and National Institute of Heart Disease, Rawalpindi, Punjab Province
  - Maryam Zahid, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Derived] Zahid M, Sughra U, Mumtaz S, Hassan M. Improving nutritional status of children using artificial intelligence-based mobile application postsurgery: randomised controlled trial. BMJ Nutr Prev Health. 2023 Dec 2;6(2):367-373. doi: 10.1136/bmjnph-2023-000645. eCollection 2023. PMID 38618548
- [Derived] Zahid M, Sughra U. Development of a protocol for conducting a randomized control trial on effects of artificial intelligence on nutritional status of children post cardiac surgery. J Pak Med Assoc. 2022 May;72(5):908-911. doi: 10.47391/JPMA.3751. PMID 35713054